CLINICAL TRIAL: NCT00002188
Title: Phase II Evaluation of Oral ALRT1057 in Patients With AIDS-Related Kaposi's Sarcoma.
Brief Title: A Study of ALRT1057 in Patients With AIDS-Related Kaposi's Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anderson Clinical Research (Industry)
Collaborators: Ligand Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 271A; L1057-28; 96ACR-LIG2
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-08

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Sarcoma, Kaposi; Antineoplastic Agents
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; AIDS-Related Opportunistic Infections | interventions — Alitretinoin

INTERVENTIONS:
Drug: Alitretinoin

SUMMARY:
The purpose of this study is to see if ALRT1057 is safe and effective in treating patients with AIDS-related Kaposi's sarcoma (KS).

DETAILED DESCRIPTION:
Patients receive open-label ALRT1057 for 16 weeks, as tolerated. In the absence of unacceptable toxicity, patients may continue treatment indefinitely provided they continue to benefit from therapy and the study remains open and active.

Thirteen patients are treated initially. If at least one response is observed in these patients, up to 14 additional patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV positive status and histologic confirmation of KS.
* CD4 count > 200 mm3 (required of one-half of patients).
* Minimum of 6 mucocutaneous KS lesions, including at least 3 raised lesions meeting criteria for "indicator" lesions.
* Acceptable organ system function.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

Serious or intercurrent illness or infection that would interfere with the ability of the patient to carry out the treatment program.

Prior Medication:

Excluded:

* Systemic therapy for KS within 30 days.
* Local or topical therapy for KS indicative lesions within 60 days.
* Systemic therapy with vitamin A in doses exceeding 15,000 IU per day or other retinoid class drug.

Required:

Approved antiretroviral therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27